CLINICAL TRIAL: NCT05606653
Title: Physiological Study of the Critical Closing Airway Pressure in a Population of Didgeridoo Players
Acronym: SASDICrit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: APHP210532
Record Dates: First submitted 2022-10-31; First posted 2022-11-07 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Sleep Apnea Syndromes
Keywords: sleep apnea syndrome; didgeridoo; uper airway
MeSH Terms: conditions — Sleep Apnea Syndromes | interventions — Respiratory Physiological Phenomena

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- didgeridoo players (Other): subjects having a regular practice of didgeridoo
  Interventions: Other: Measurement of critical airway closing pressure; Other: Respiratory function tests; Other: pharyngometry
- oboe players (Other): subjects having a regular practice of the oboe
  Interventions: Other: Measurement of critical airway closing pressure; Other: Respiratory function tests; Other: pharyngometry
- control (Other): control subjects without diagnosed SAS, at low risk of SAS on the Berlin questionnaire and the STOP BANG questionnaire
  Interventions: Other: Measurement of critical airway closing pressure; Other: Respiratory function tests; Other: pharyngometry

INTERVENTIONS:
Other: Measurement of critical airway closing pressure — Measurement of critical airway closing pressure
Other: Respiratory function tests — CO2 response test
Other: pharyngometry — measure of the pharyngometry

SUMMARY:
Obstructive sleep apnea is characterised by an abnormal upper airway collapsibility. Upper airway collapsibility can be evaluated through critical closure airway pressure (Pcrit). Didgeridoo is a traditional australian musical instrument involving circular respiration, a breathing technique involving mouth muscles. We hypothesize that didgeridoo players have a lower risk of airway collapsibility due to circular breathing technique

DETAILED DESCRIPTION:
Some studies have shown the benefit of playing the didgeridoo, a wind musical instrument of Aboriginal origin, on the risk of obstructive sleep apnea hypopnea syndrome (OSAHS) and on OSAHS itself. Thus, didgeridoo players are less at risk of OSAHS and the practice of this instrument reduces the severity of this syndrome. To date, there are very few studies on the physiological mechanisms involved in the practice of the didgeridoo to explain this reduction in risk and impact on OSAHS.

The rare studies carried out show a great participation of the dilator muscles of the pharynx. We can also note that the didgeridoo is practiced with a particular breathing technique allowing air to be expelled while inhaling. This technique is called circular breathing. This breathing is acquired by working on the control of these dilator muscles of the pharynx but also by becoming aware of its ventilatory needs. Thus it is for the players to learn to breathe according to the needs without disturbing the piece. This respiratory learning, ventilation modulation, not explored until now, could influence the sensitivity of the central and peripheral chemoreceptors of the player with respect to his pCO2 and his pO2. We know the role of this sensitivity in the pathophysiology of SAS.

In this work we therefore seek to highlight a benefit to the practice of the didgeridoo on the critical pressure of pharyngeal closure involving the dilator muscles of the pharynx but also a benefit in terms of gas exchange by analyzing the slope of response to CO2 .

We will compare the effect of using the didgeridoo with that of another wind instrument, the oboe, on these respiratory parameters.

We chose this instrument because a study showed a lower risk of SAS in a population of oboe players. However, in the practice of this instrument, circular breathing is not used.

It would therefore be a comparative observational study with the recruitment of three groups of subjects in order to:

* Compare didgeridoo players with subjects not playing a wind instrument;
* Compare didgeridoo players with players of another wind instrument. There is no fixed reference value for Pcrit in healthy subjects, partly due to the heterogeneity of VAS collapsibility in healthy subjects (Pcrit is between -5 and -25 cm d water according to the studies), and on the other hand the wide variety of measurement methods. It is therefore necessary to have control groups.

Given the epidemiology of obstructive SAS and the exploratory nature of this study, we decided to include only male subjects, which will also make it possible to eliminate the effects of sex on respiratory chemosensitivity. Similarly, given the epidemiology of SAS, an age limit of 85 years was introduced in order not to overlook the effects of aging on the collapsibility of the VAS and chemosensitivity.

Finally, subjects will be matched on age (+/- 5 years) and body mass index (BMI, +/- 2.5 kg/m2) as there is a relationship between age/BMI and the collapsibility of the VAS on the one hand, and between age/BMI and the occurrence of SAS on the other hand.

"

ELIGIBILITY:
Inclusion criteria :

* Male patient
* Age ≥18 and ≤85 years old
* Free, informed and written consent
* Affiliation to a social security scheme

For "Didgeridoo players" group:

- Regular practice of the didgeridoo defined by a practice of more than 3 times a week, for more than 1 year and having acquired the circular breathing technique.

For "Oboe players" group:

- Regular practice of the oboe defined by a practice of more than 3 sessions per week for more than 1 year.

For "Control cases" group:

- Patient free from SAS and at low risk of SAS on the Berlin questionnaire and the STOP BANG questionnaire.

Exclusion criteria :

* Participation in a research protocol involving the human person in the previous months if an exclusion instruction is given in this protocol
* Use of respiratory depressants or sedatives, systemic corticosteroid therapy
* Unstable cardiovascular disease (cardiovascular event less than a month old)
* Recent ENT surgery (less than 6 months)
* Known central neurological pathology
* Psychiatric pathology according to DSM-V criteria, unbalanced
* Pulsed oxyhemoglobin saturation < 88% at rest, while awake
* Patient under guardianship or curators
* Patient under AME
* Absence of prior medical examination"

Ages: 18 Years to 85 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2021-09-16 (Actual); Primary Completion 2023-07-07 (Actual); Study Completion 2024-01-16 (Actual)

PRIMARY OUTCOMES:
values of the critical closing pressure of the VAS (Pcrit) in patients of the "Didgeridoo players" group and the "control" group | one day

SECONDARY OUTCOMES:
Value of the slope of response to CO2 in each of the three groups | one day
pharyngeal volume | one day

CONTACTS AND LOCATIONS:
Overall Officials: Frija-Masson Justine, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Justine Frija, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided